CLINICAL TRIAL: NCT06816862
Title: Clinical/Radiologic Outcomes Associated With the SYMPHONY™ OCT System for Treatment of Acute and Chronic Instabilities of the Craniocervical Junction, the Cervical Spine and the Upper Thoracic Spine
Brief Title: SYMPHONY™ OCT System for Instabilities of the Upper Thoracic and Cervical Spine
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SYMPHONY™
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cervical Instabilities Spine; Spine; Instability
Keywords: Spine Fusion; Spine Fixation; Spine Surgery; Cervical Instabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SYMPHONY™ Cohort: This cohort is composed of patients who will be prospectively enrolled (35 total). These patients will undergo upper spinal stabilisation supplemented with internal fixation using the SYMPHONY™ OCT system indicated for acute and chronic upper spinal instabilities. This device is FDA approved thus this is post market observational intervention. This trial was a target follow up of 2 years for each participant.
  Interventions: Device: SYMPHONY™ OCT System

INTERVENTIONS:
Device: SYMPHONY™ OCT System — Internal fixation system for surgical stabilisation of upper spine instabilities

SUMMARY:
This will be a prospective, multi-centre study at a National Tertiary Referral Centre for spinal trauma and spinal cord injuries, serving a catchment area of 5 million people. Consecutive patients undergoing posterior-only surgery or combined anterior and posterior surgery for degenerative cervical pathology, traumatic spinal fractures or dislocations, failed previous fusions or treatment for tumour involving the cervical/thoracic spine will be enrolled. This is a post-market trial, with a CE-marked medical device called the SYMPHONY OCT System which is currently in use in both centres. The SYMPHONY™ OCT System is a portfolio of internal fixation tools including screw, rods and hooks used as an adjunct to fusion for posterior stabilisation of the upper spine in skeletally mature patients. This pilot study hypothesizes that the use of SYMPHONY™ OCT System to treat upper spine instabilities will achieve results comparable to historical cases using the Mountaineer performed until 2021.

DETAILED DESCRIPTION:
This will be a prospective, multi-centre study at a National Tertiary Referral Centre for spinal trauma and spinal cord injuries, serving a catchment area of 5 million people. This study will follow patients undergoing posterior stabilisation of the upper spine using the SYMPHONY™ OCT system as an augment to fusion. This system consists of bone anchors (e.g. screws) for connection by longitudinal components (e.g. rods) via an interconnection mechanism (e.g., set screws) with optional transverse connectors (e.g., cross connectors) to link longitudinal components for additional stability during fusion mass development.

In spine fusion procedures, bone is encouraged to grow in order to fuse vertebrae of the spine together to relieve pain or increase stability. The likelihood of a successful fusion is thought to be influenced by multiple factors. Patient-related factors influencing fusion success include comorbidities such as osteoporosis or osteopenia, diabetes, and obesity. Factors affecting the inflammatory response, such as rheumatoid arthritis or long-term steroid use may also increase the likelihood of fusion failure. Fusion success can also be influenced by age, frailty, functional status, history of smoking or steroid use.

Frailty is a clinically recognizable syndrome comprised of declining physiological reserve, characterized by decreased resilience to adverse health outcomes. Fried et al have defined frailty as meeting three out of five of the following criteria: low grip strength, low energy, slow walking speed, low physical activity, unintentional weight loss. The modified 5-item frailty index (mFI-5) is another method of measuring frailty commonly used in clinical settings. It has been shown to predict the occurrence of adverse outcomes following various orthopaedic surgeries. The five comorbidities included in the mFI-5 are a history of hypertension, COPD, diabetes mellitus, congestive heart failure, and a non-independent functional status.

This pilot study hypothesizes that the use of SYMPHONY™ OCT System to treat upper spine instabilities will achieve results comparable to historical cases using the Mountaineer performed until 2021.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients presenting for the treatment of acute and chronic instabilities of the craniocervical junction, the cervical and upper thoracic spine for whom the SYMPHONY OCT System is a suitable choice will be included in this study.
* Patients undergoing surgical treatment for upper cervical spine traumatic spinal fractures and/or traumatic dislocations, failed previous fusions (pseudarthrosis) and tumours involving the cervical/thoracic spine will be included in this study.

Exclusion Criteria:

* Non-surgical candidates, patients with contraindications to surgery (e.g. severe medical comorbidities, known infection, etc.),
* Patients with established osteoporosis
* Long-term, systemic steroid use
* Systemic diseases (e.g. rheumatoid arthritis, AIDS, HIV, etc.),
* Patients unwilling or unable to give informed consent, or patients unwilling or unable to complete Health-related quality of (HRQOL) outcome life measures at the specified study time points pre- and post-operatively.
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years or older) with acute/chronic upper spine instabilities requiring surgical intervention and stabilisation with instrumentation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion at 24 months as inferred by Presence of Segmental Stability and Absence of Mechanical Failure on Xray/CT | 24 months
  The primary objective of this study is to evaluate the radiographic assessment of fusion at 24 months postoperatively. This radiographic assessment will consist of plain Xrays preoperatively, at 6 weeks, 3 months, 6 months and 24 months postoperatively. These will include a combination of anterior, lateral, flexion and extension views images of the spine used to infer stability.
  Fusion failure (pseudarthrosis) will be defined as signs of mechanical failure (such as peri-implant radiolucency/haloing, screw/rod fracture, etc.) or <50% bridging trabecular bone on CT scan at 12 months postoperatively. Assessment of fusion will be conducted by a musculoskeletal radiologist and 2 independent fellowship trained spine surgeons.

SECONDARY OUTCOMES:
Changes in Patient Reported Pain as Measured Using Visual Analogue Scale Score Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient pain will be recorded using the Visual Analogue Scale which ranges from 0 to 10 with a score of 10 indicating the most severe possible pain and a score of 0 indicating no pain is present.
  A secondary objective of this study is to prospectively gather patient reported outcomes (PROMs) in terms of pain and function
Changes in Patient Reported Function as Measured Using Short Form 12 Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient function will be recorded using the Short Form 12 which returns component scores representing both physical and mental status. These scores are adjusted and compare versus averages within the United States population. Both scores have an average score of 50 with a standard deviation of 10. Lower scores indicate worse function while higher scores indicate greater function.
Changes in Patient Reported Function as Measured Using Neck Disability Index Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient function will be recorded using the Neck Disability Index which ranges from 0 to 100 disability with a score of 100% indicating complete disability and a score of 0% indicating no disability is present.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Butler, PhD, Principal Investigator — Mater Misericordiae University Hospital
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No
Analysis / breakdown of IPD is not felt to benefit study results or outcomes based on the study methodology.

REFERENCES:
- [Background] Verla T, Xu DS, Davis MJ, Reece EM, Kelly M, Nunez M, Winocour SJ, Ropper AE. Failure in Cervical Spinal Fusion and Current Management Modalities. Semin Plast Surg. 2021 Feb;35(1):10-13. doi: 10.1055/s-0041-1722853. Epub 2021 May 10. PMID 33994872
- [Background] Badiee RK, Mayer R, Pennicooke B, Chou D, Mummaneni PV, Tan LA. Complications following posterior cervical decompression and fusion: a review of incidence, risk factors, and prevention strategies. J Spine Surg. 2020 Mar;6(1):323-333. doi: 10.21037/jss.2019.11.01. PMID 32309669
- [Background] Hilibrand AS, Fye MA, Emery SE, Palumbo MA, Bohlman HH. Impact of smoking on the outcome of anterior cervical arthrodesis with interbody or strut-grafting. J Bone Joint Surg Am. 2001 May;83(5):668-73. doi: 10.2106/00004623-200105000-00004. PMID 11379735
- [Background] Lau D, Chou D, Ziewacz JE, Mummaneni PV. The effects of smoking on perioperative outcomes and pseudarthrosis following anterior cervical corpectomy: Clinical article. J Neurosurg Spine. 2014 Oct;21(4):547-58. doi: 10.3171/2014.6.SPINE13762. Epub 2014 Jul 11. PMID 25014499
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Platt D, Platt M, Loffler H. [Cytochemical demonstration of beta-acetylglucosamindase in human blood- and bone marrow cells]. Klin Wochenschr. 1968 Jun 1;46(11):617-8. doi: 10.1007/BF01747843. No abstract available. German. PMID 5726589